CLINICAL TRIAL: NCT01393795
Title: A Double-blind, Randomized, Crossover Clinical Study to Assess the Efficacy of Qutenza® for the Reduction of Site Pain Caused by Continuous Subcutaneous Infusion of Remodulin®, in Pulmonary Arterial Hypertension Patients
Brief Title: Qutenza®-Remodulin® in Pulmonary Arterial Hypertension Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO1824
Record Dates: First submitted 2011-06-22; First posted 2011-07-13 (Estimated); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Hypertension; Pain
Keywords: Pulmonary Hypertension; Pain
MeSH Terms: conditions — Hypertension, Pulmonary; Pain | interventions — Capsaicin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tegaderm (Placebo Comparator)
  Interventions: Drug: Tegaderm
- Qutenza (Active Comparator)
  Interventions: Drug: Qutenza

INTERVENTIONS:
Drug: Qutenza — 8% patch
  Arms: Qutenza
Drug: Tegaderm — No active drug
  Arms: Tegaderm

SUMMARY:
The investigators hypothesise that pre-application of Qutenza® patches to the skin may reduce pain at the site of Remodulin® SC infusion (sited 1 to 2 weeks later at the site of Qutenza pre-application), in which case it would greatly improve the quality of life of the patients, and enable many more to continue with this treatment. It may also provide new information to support the use of Qutenza® patches for preventing and reducing pain produced by inflammation.

The present study will explore the efficacy of single applications of Qutenza® (capsaicin 8% patch) in reducing site pain caused by continuous SC infusion of Remodulin®, in pulmonary arterial hypertension patients, as assessed by changes in subjective pain rating score and/or pain and sensory testing.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older with symptomatic PAH
* Willing to provide written informed consent to participate in the study.
* With documented diagnosis of PAH, either idiopathic, familial or associated with connective tissue disease, congenital heart disease or the use of anorexogenic drugs.
* Documented haemodynamic diagnosis of PAH by right heart catheterization - performed at any time prior to screening, showing: mean pulmonary arterial pressure >25 mm Hg, pulmonary capillary wedge pressure =/< 15 mmHg and pulmonary vascular resistance >240 dynes/sec/cm
* Receiving stable doses of Remodulin® SC, continuously infused at a dose of at least 2.5 ng/kg/min for at least 8 weeks prior to enrolment. Additional medications that are approved for treatment of PAH (either bosentan or sildenafil) and other supplementary treatments such as oral anticoagulants, diuretics, digitalis, calcium channel blockers or oxygen supplementation are permitted.
* History of pain at the site of Remodulin® SC infusion for at least 8 weeks prior to enrolment and as assessed on the 11 point pain intensity numerical pain rating scale (NPRS) from 0 to 10, where 0 represents "No pain" and 10 represents "Maximum pain imaginable". Patients with a history of pain intensity equal or greater than 3 NPRS points (as determined by the NPRS trial diary completed during the screening period) are eligible to participate.
* Modified New York Heart Association (NYHA) (WHO) classification II-IV that has been stable for at least 8 weeks prior to enrolment.
* A female subject is eligible to participate if she is of:

  * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol <40 pg/ml (<140 pmol/L) is confirmatory].
  * Child-bearing potential and agrees to use one of the contraception methods listed in the protocol.

Exclusion Criteria:

* Patient's participating in another clinical trial or who have done so within 30 days before screening.
* Patients with PAH in NYHA/WHO functional class I at screening.
* Known to be positive for human immunodeficiency virus (HIV).
* Patients with any additional medical condition or illness that, in the opinion of the Investigator would interfere with study compliance and/or impair the patient's ability to participate or complete the study.
* Patients with a history of substance abuse (e.g. alcohol or drug abuse) within the previous 6 months before enrolment.
* Patients with a history of severe allergies or multiple drug allergies and/or reported hypersensitivity to capsaicin.
* Patients with no history of pain at the site of Remodulin® SC infusion or average pain intensity at screening less than 3 points on the numerical pain rating scale (NPRS).
* Life expectancy less than 12 months.
* Unable to provide informed consent.
* Female patients who are lactating or pregnant (positive pre-randomisation serum pregnancy test) or plan to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Safety Measures | Approximately 9 months (vital signs, AE's and concomitant medications will be recorded throughout the study)
  Safety evaluations will be based on the incidence, intensity and type of AEs and clinically significant changes in vital signs (pulse rate, blood pressure, respiration rate, pulse oximetry and temperature), and changes in concomitant medications throughout the study.
  Evaluation of safety will also be based on subject's physical examination, signs and symptoms of PAH, routine clinical laboratory tests (hematology, chemistry, coagulation panel, and urinalysis), ECG, and NYHA (WHO) classification at the screening and end of study follow up visits.

SECONDARY OUTCOMES:
Efficacy measure - change in mean NPRS score | Approximately 9 months. Average daily NPRS scores from Weeks 1 and 2 of each treatment period will be expressed as percentage changes from the average daily NPRS score at baseline
  The primary efficacy measure will be the change in mean NPRS pain score (reduced by greater than 1.1) at the site of Remodulin® SC infusion, following Qutenza® or transparent adhesive control dressing (Tegaderm film 10cmx12cm) in combination with 0.075% capsaicin cream (Axsain®), during two treatment periods. Efficacy of Qutenza® relative to the control will also be assessed on PGIC, as well as sensory tests and flare area.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Libri, MD, Principal Investigator — Imperial College London
Locations (1):
- Hammersmith Hospital, Imperial College NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Libri V, Gibbs JS, Pinato DJ, Iddamalgoda T, Khengar RH, Gin-Sing W, Huson L, Anand P. Capsaicin 8% patch for treprostinil subcutaneous infusion site pain in pulmonary hypertension patients. Br J Anaesth. 2014 Feb;112(2):337-47. doi: 10.1093/bja/aet308. Epub 2013 Sep 22. PMID 24062200